CLINICAL TRIAL: NCT05937282
Title: Comparative Study Between the Hemodynamic Responses of Dexmedetomidine, Lidocaine or Propofol Infusions During Laparoscopic Cholecystectomy
Brief Title: Hemodynamic Responses of Dexmedetomidine, Lidocaine or Propofol Infusions During Laparoscopic Cholecystectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Nasar, Specialist, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2/2020ANET27
Record Dates: First submitted 2023-06-18; First posted 2023-07-10 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Hemodynamic Responses; Laparoscopic Cholecystectomy; Dexmedetomidine; Lidocaine; Propofol
MeSH Terms: interventions — Dexmedetomidine; Propofol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Control group (Placebo Comparator): Patients will receive infusion of 25 ml normal saline in 50 ml syringe pump.
  Interventions: Drug: normal saline
- Dexmedetomidine group (Active Comparator): Patients will receive infusion of dexmedetomidine in the dose of 0.4 μg/kg/hr. One ml dexmedetomidine (100 μg/ml) will be diluted with 24 ml normal saline in 50 ml syringe pump to achieve dilution of 4 μg/ml.
  Interventions: Drug: Dexmedetomidine
- Propofol (Active Comparator): Patients will receive propofol infusion in the dose of 3 mg/kg/hr. (12) 25 ml propofol 1% (10 mg /ml) in 50 ml syringe pump
  Interventions: Drug: Propofol
- Lidocaine (Active Comparator): Patients will receive lidocaine infusion in the dose of 2 mg /kg/hr. (15) 25 ml lidocaine 1% (10 mg/ml) in 50 ml syringe pump.
  Interventions: Drug: Lidocain

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will receive infusion of dexmedetomidine in the dose of 0.4 μg/kg/hr. One ml dexmedetomidine (100 μg/ml) will be diluted with 24 ml normal saline in 50 ml syringe pump to achieve dilution of 4 μg/ml.
  Arms: Dexmedetomidine group
Drug: Propofol — Patients will receive propofol infusion in the dose of 3 mg/kg/hr. 25 ml propofol 1% (10 mg /ml) in 50 ml syringe pump.
  Arms: Propofol
Drug: Lidocain — Patients will receive lidocaine infusion in the dose of 2 mg /kg/hr.25 ml lidocaine 1% (10 mg/ml) in 50 ml syringe pump.
  Arms: Lidocaine
Drug: normal saline — Patients will receive infusion of 25 ml normal saline in 50ml syringe pump (control group).
  Arms: Control group

SUMMARY:
This study will be carried out to compare the efficacy of dexmedetomidine, propofol or lidocaine infusions in attenuation of hemodynamic responses to pneumoperitoneum during adult laparoscopic cholecystectomy using electrical cardiometry.

DETAILED DESCRIPTION:
Many drug infusions have been used to control hemodynamic responses to laparoscopic surgeries like propofol, fentanyl, esmolol with varying degrees of success.

Dexmedetomidine has sedative and analgesic properties seems to be appropriate enough to control the sympathetic response as well as provide a stable hemodynamics

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists I patients.
* Patients between the ages of ≥ 20 and ≤ 60 years of both sexes.

Exclusion Criteria:

* Hypersensitivity to dexmedetomidine, propofol or lidocaine.
* Diabetic patients (Hemoglobin A1C ≥ 7).
* Hypertensive patients (Blood presssure ≥ 140/90 mmHg) or patients on medications that affect hemodynamics as clonidine, methyldopa, β blockers and calcium channel blockers.
* Impaired liver function (serum albumin ≤ 3.5 g/dl, International normalized ratio≥ 1.3, total bilirubin >1mg/dl).
* Impaired renal function (serum creatinine >1.2 mg/dl, blood urea >20mg/dl).
* Morbidly obese patients with body mass index ≥ 40.
* Patients with acute cholecystitis or active infection.
* Patients taking medications that may impair cognition.
* History of seizures.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Noninvasive mean blood pressure | Intraoperatively
  mean blood pressure will be noted by a standard automated multi channel monitor will be connected to each patient

SECONDARY OUTCOMES:
Intraoperative rescue drugs | Intraoperatively
  Patients that will need rescue drugs (fentanyl) will be recorded with the total dose used.
Post extubation sedation | 24 hour postoperatively
  Post extubation sedation assessment will be done in each group using Ramsey's sedation score.
  Anxious, agitated or restless = (1) Cooperative, oriented and tranquil = (2) Responsive to command only = (3) Brisk response to light glabellar tap or loud auditory stimulus = (4) Sluggish response to light glabellar tap or loud auditory stimulus = (5) No response = (6)

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia University, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the corresponding author from one year after study completion
Time Frame: from one year after study completion
Access Criteria: The data will be available upon reasonable request from the corresponding author